CLINICAL TRIAL: NCT06780501
Title: Neuropsychiatric Research Databases for People With Intellectual Disabilities and Epilepsy (REFINE)
Acronym: REFINE
Status: Recruiting | Type: Observational
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Professor Rohit Shankar, Professor in Neuropsychiatry, University of Plymouth
Other Study IDs: 5284
Record Dates: First submitted 2024-09-19; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-09

CONDITIONS: Epilepsy; Intellectual Disability; Learning Disability
MeSH Terms: conditions — Epilepsy; Intellectual Disability; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study consists of two parts:

Part One: De-identified Database

The goal of this part is to establish a research database containing de-identified data about People with Intellectual Disabilities (PwID) and epilepsy, collected from three NHS sites across England and Wales. Researchers will gather information from participants' medical records, including clinical details, epilepsy history, and medications, and will enter this data into a secure database where all identifying details are removed. This part of the study aims to determine whether it's possible to identify eligible participants, collect complete datasets for each participant, and identify any issues that may affect the quantity and quality of data. These findings will help inform a potential future study that could involve 20 or more sites.

Part Two: Research Register

The goal of this part is to create a research register of individuals with PwID and epilepsy. Participants will be approached and asked for their consent to collect their personal and clinical data, which will help identify those willing to take part in future ethically approved research projects. As in Part One, researchers will collect data from medical records. Participants who consent to be included in the register may be contacted by external researchers for future studies. The aim is to facilitate national collaboration by enabling data sharing between research projects, thereby improving the ability to answer more questions and enhance patient care. This part of the study will test whether it's possible to determine screening and recruitment rates at each site, develop and evaluate recruitment processes, and assess how researchers leading other approved studies can obtain permission to use the register. Additionally, it will evaluate whether it's possible to collect a complete dataset for each participant.

ELIGIBILITY:
The de-identified database:

Inclusion Criteria:

* Clinical diagnosis of ID in medical records.
* Clinical diagnosis of epilepsy in medical records.
* Patient is over the age of 18 years old.
* Under the current care of specialist ID or epilepsy services at one of the three participating NHS Trusts.

Exclusion Criteria:

* Other neurodevelopmental disorders without ID.
* Patient is recorded on the National Data Opt-out as not wishing their data to be used for research/audit.

The research register:

Inclusion Criteria:

* Clinical diagnosis of ID in medical records.
* Clinical diagnosis of epilepsy in medical records.
* Under the current care of specialist ID or epilepsy services at one of the three participating NHS Trusts.
* Between the ages of 18 and 30 at the time of consent.
* Participant has the capacity to be able to provide consent for themselves, or a personal consultee is able to provide an opinion on the views and feelings of the potential participant.
* Patients (or personal consultee) must be able to communicate in English (or Welsh in Welsh site).

Exclusion Criteria:

- Other neurodevelopmental disorders without ID.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a clinical diagnosis of an Intellectual Disability (ID) and epilepsy at participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The set up of a research database consisting of de-identified data focused on People with Intellectual Disabilities (PwID) and epilepsy at three UK NHS sites across England and Wales. | End of study (May 2025)
  De-identified database
The development of a research register of PwID and epilepsy. Participants will consent to the collection of their personal/clinical data, which will enable the identification of patients willing to take part in other ethically approved research projects. | End of study (May 2025)
  Research register

SECONDARY OUTCOMES:
Numbers of eligible patients identified at each site for data collection (De-identified database). | End of study (May 2025)
  Feasibility objective
Completeness of clinical data collected (De-identified database) | End of study (May 2025)
  Feasibility objective
Feedback collected from sites about any issues around identifying patients and locating the data required (De-identified database). | End of study (May 2025)
  Feasibility objective
Screening and recruitment rates at each site (Research register). | End of study (May 2025)
  Feasibility objective
Successful recruitment process in place at each site (Research register). | End of study (May 2025)
  Feasibility objective
Set up of a formal process including the REFINE Study Oversight Committee to review requests for access to the participant register (Research register). | End of study (May 2025)
  Feasibility objective
Completeness of clinical data collected (Research register). | End of study (May 2025)
  Feasibility objective

CONTACTS AND LOCATIONS:
Overall Officials: Lance Watkins, Principal Investigator — Swansea Bay University Health Board; Sarah Lennard, Principal Investigator — Cornwall Partnership NHS Foundation Trust; Heather Angus-Leppan, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Cornwall Partnership NHS Foundation Trust, Bodmin
  - Royal Free London Hospitals NHS Trust, London
  - Swansea Bay University Health Board, Swansea

REFERENCES:
- [Derived] Musicha C, Neilens H, Stanyard E, Allgar V, Lomax J, Ashford R, Hambly H, Aspinall P, O'Shaughnessy E, Rollinson C, Lennard S, Mclean B, Simpson A, Bowman P, Angus-Leppan H, Watkins L, Laugharne R, Allard J, Shankar R. Neuropsychiatric research databases for people with intellectual disabilities and epilepsy (REFINE): a feasibility study protocol. BMJ Open. 2025 Nov 26;15(11):e108869. doi: 10.1136/bmjopen-2025-108869. PMID 41298255